CLINICAL TRIAL: NCT00983853
Title: A Phase 2a, 2-Part, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study of Telaprevir in Combination With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Subjects Who Have Chronic HCV-1/HIV-1 Co-Infection and Are Treatment-Naïve for Hepatitis C
Brief Title: Safety and Efficacy of Telaprevir in Combination With Peginterferon Alfa-2a and Ribavirin in Subjects Co-Infected With Hepatitis C Virus (HCV) and HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX08-950-110
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C; HIV Infections
Keywords: VX-950; INCIVEK; INCIVO
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): The dose of ribavirin used (fixed versus weight-based) is region dependent
  Interventions: Drug: telaprevir or matching placebo; Biological: peginterferon alfa-2a; Drug: ribavirin (fixed dose); Drug: ribavirin (weight-based dose)
- Part B (Experimental): The dose of ribavirin used (fixed versus weight-based) is region dependent
  Interventions: Drug: telaprevir or matching placebo; Biological: peginterferon alfa-2a; Drug: ribavirin (fixed dose); Drug: ribavirin (weight-based dose)

INTERVENTIONS:
Drug: telaprevir or matching placebo — Tablet, Oral, 750 mg, q8h, 12 weeks
  Arms: Part A
Drug: telaprevir or matching placebo — Tablet, Oral, 750 mg or 1125 mg, q8h, 12 weeks
  Arms: Part B
Biological: peginterferon alfa-2a — Subcutaneous injection, 180 μg, once weekly, 48 weeks
Drug: ribavirin (fixed dose) — Tablet, Oral, 800 mg, b.i.d., 48 weeks
Drug: ribavirin (weight-based dose) — Tablet, Oral, 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d., 48 weeks

SUMMARY:
The purpose of this study is to determine whether the combination of telaprevir, peginterferon alfa-2a, and ribavirin is safe and effective in treating hepatitis C virus (HCV) infection in subjects who are infected with both HCV and human immunodeficiency virus (HIV).

ELIGIBILITY:
Inclusion Criteria:

* Chronic, genotype 1, hepatitis C with detectable HCV RNA
* HIV-1 infection for >6 months
* Documentation of a liver biopsy within 1 year before the screening visit showing evidence of hepatitis (demonstrated by inflammation and/or fibrosis)

Exclusion Criteria:

* Previous treatment with any approved or investigational drug or drug regimen for the treatment of hepatitis C
* Previous treatment with interferon or ribavirin
* Evidence of hepatic decompensation in cirrhotic subjects
* Subjects who have participated in a clinical study involving administration of an investigational drug within 2 months
* Part A only: subjects who have been on a HAART regimen within 12 weeks before study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (16):
- United States (11):
  - Beverly Hills, California
  - San Diego, California
  - San Francisco, California
  - Miami, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Cincinnati, Ohio
  - Dallas, Texas
- Paris, France
- Germany (2):
  - Bonn-Venusberg
  - Hamburg
- Spain (2):
  - Barcelona
  - Madrid

REFERENCES:
- [Derived] Sulkowski MS, Sherman KE, Dieterich DT, Bsharat M, Mahnke L, Rockstroh JK, Gharakhanian S, McCallister S, Henshaw J, Girard PM, Adiwijaya B, Garg V, Rubin RA, Adda N, Soriano V. Combination therapy with telaprevir for chronic hepatitis C virus genotype 1 infection in patients with HIV: a randomized trial. Ann Intern Med. 2013 Jul 16;159(2):86-96. doi: 10.7326/0003-4819-159-2-201307160-00654. PMID 23685940

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: T/PR: Drug: telaprevir tablet, oral, 750 mg, q8h, 12 weeks
  Biological: peginterferon alfa-2a subcutaneous injection, 180 μg, once weekly, 48 weeks
  Drug: ribavirin (fixed dose) tablet, oral, 800 mg, b.i.d., 48 weeks
  Drug: ribavirin (weight-based dose) tablet, oral, 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d., 48 weeks
  The dose of ribavirin used (fixed versus weight-based) was region dependent.
- Part A: Pbo/PR: Drug: placebo tablet, oral, 750 mg, q8h, 12 weeks
  Biological: peginterferon alfa-2a subcutaneous injection, 180 μg, once weekly, 48 weeks
  Drug: ribavirin (fixed dose) tablet, oral, 800 mg, b.i.d., 48 weeks
  Drug: ribavirin (weight-based dose) tablet, oral, 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d., 48 weeks
  The dose of ribavirin used (fixed versus weight-based) was region dependent.
- Part B: EFV-based HAART + T/PR: Drug: efavirenz, tenofovir disoproxil fumarate, and emtricitabine
  Drug: telaprevir tablet, oral, 750 mg, q8h, 12 weeks
  Biological: peginterferon alfa-2a subcutaneous injection, 180 μg, once weekly, 48 weeks
  Drug: ribavirin (fixed dose) tablet, oral, 800 mg, b.i.d., 48 weeks
  Drug: ribavirin (weight-based dose) tablet, oral, 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d., 48 weeks
  The dose of ribavirin used (fixed versus weight-based) was region dependent.
- Part B: EFV-based HAART + Pbo/PR: Drug: efavirenz, tenofovir disoproxil fumarate, and emtricitabine
  Drug: placebo tablet, oral, 750 mg, q8h, 12 weeks
  Biological: peginterferon alfa-2a subcutaneous injection, 180 μg, once weekly, 48 weeks
  Drug: ribavirin (fixed dose) tablet, oral, 800 mg, b.i.d., 48 weeks
  Drug: ribavirin (weight-based dose) tablet, oral, 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d., 48 weeks
  The dose of ribavirin used (fixed versus weight-based) was region dependent.
- Part B: ATV/R-based HAART + T/PR: Drug: ritonavir-boosted atazanavir, tenofovir disoproxil fumarate, and emtricitabine or lamivudine
  Drug: telaprevir tablet, oral, 750 mg, q8h, 12 weeks
  Biological: peginterferon alfa-2a subcutaneous injection, 180 μg, once weekly, 48 weeks
  Drug: ribavirin (fixed dose) tablet, oral, 800 mg, b.i.d., 48 weeks
  Drug: ribavirin (weight-based dose) tablet, oral, 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d., 48 weeks
  The dose of ribavirin used (fixed versus weight-based) was region dependent.
- Part B: ATV/R-based HAART + Pbo/PR: Drug: ritonavir-boosted atazanavir, tenofovir disoproxil fumarate, and emtricitabine or lamivudine
  Drug: placebo tablet, oral, 750 mg, q8h, 12 weeks
  Biological: peginterferon alfa-2a subcutaneous injection, 180 μg, once weekly, 48 weeks
  Drug: ribavirin (fixed dose) tablet, oral, 800 mg, b.i.d., 48 weeks
  Drug: ribavirin (weight-based dose) tablet, oral, 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d., 48 weeks
  The dose of ribavirin used (fixed versus weight-based) was region dependent.
Period: Overall Study
Arm/Group | Part A: T/PR | Part A: Pbo/PR | Part B: EFV-based HAART + T/PR | Part B: EFV-based HAART + Pbo/PR | Part B: ATV/R-based HAART + T/PR | Part B: ATV/R-based HAART + Pbo/PR
Started | 7 | 7 (1 subject was randomized but not dosed) | 17 (1 subject was randomized but not dosed) | 8 | 15 | 8
Completed | 6 | 5 | 14 | 6 | 12 | 7
Not Completed | 1 | 2 | 3 | 2 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Unable to come to study follow-up visits | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least 1 dose of study drug
Groups:
- Part A: T/PR: Telaprevir plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects not receiving HAART.
- Part A: Pbo/PR: Placebo plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects not receiving HAART.
- Part B: EFV-based HAART + T/PR: Telaprevir plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant efavirenz(EFV)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
- Part B: EFV-based HAART + Pbo/PR: Placebo plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant efavirenz(EFV)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
- Part B: ATV/R-based HAART + T/PR: Telaprevir plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant ritonavir-boosted atazanavir(ATV/r)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
- Part B: ATV/R-based HAART + Pbo/PR: Placebo plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant ritonavir-boosted atazanavir(ATV/r)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
- Total: Total of all reporting groups
Arm/Group | Part A: T/PR | Part A: Pbo/PR | Part B: EFV-based HAART + T/PR | Part B: EFV-based HAART + Pbo/PR | Part B: ATV/R-based HAART + T/PR | Part B: ATV/R-based HAART + Pbo/PR | Total
Number analyzed (Participants) | 7 | 6 | 16 | 8 | 15 | 8 | 60
Age Continuous [Median (Full Range); unit: years]
  median (min, max) | 39.4 [34 to 50] | 47.5 [42 to 65] | 47.5 [31 to 57] | 47.0 [31 to 53] | 52.0 [36 to 59] | 39.0 [26 to 53] | 44.5 [26 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 | 2 | 1 | 7
  Male | 6 | 4 | 16 | 7 | 13 | 7 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5 | 1 | 3 | 3 | 17
  Not Hispanic or Latino | 4 | 4 | 10 | 7 | 12 | 5 | 42
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2 | 3 | 12 | 5 | 13 | 7 | 42
  Black/African American | 4 | 3 | 3 | 3 | 2 | 1 | 16
  American Indian/Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  North America | 7 | 5 | 13 | 8 | 9 | 4 | 46
  United States | 7 | 5 | 13 | 8 | 9 | 4 | 46
  Europe | 0 | 1 | 3 | 0 | 6 | 4 | 14
  Germany | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Spain | 0 | 1 | 2 | 0 | 3 | 3 | 9
  France | 0 | 0 | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Undetectable HCV RNA at Week 12
Time Frame: 12 weeks after first dose of study drug
Population: Subjects who were randomized and received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Part B: EFV-based HAART + T/PR: Telaprevir plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant efavirenz (EFV)-based highly active antiretroviral therapy (HAART) for the entire 48 week study.
- Part B: EFV-based HAART + Pbo/PR: Placebo plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant efavirenz (EFV)-based highly active antiretroviral therapy (HAART) for the entire 48 week study.
- Part B: ATV/R-based HAART + T/PR: Telaprevir plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant ritonavir-boosted atazanavir (ATV/r)-based highly active antiretroviral therapy (HAART) for the entire 48 week study.
- Part B: ATV/R-based HAART + Pbo/PR: Placebo plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant ritonavir-boosted atazanavir (ATV/r)-based highly active antiretroviral therapy (HAART) for the entire 48 week study.
Arm/Group | Part A: T/PR | Part A: Pbo/PR | Part B: EFV-based HAART + T/PR | Part B: EFV-based HAART + Pbo/PR | Part B: ATV/R-based HAART + T/PR | Part B: ATV/R-based HAART + Pbo/PR
Number analyzed (Participants) | 7 | 6 | 16 | 8 | 15 | 8
participants | 6 | 2 | 14 | 2 | 10 | 2

2. Secondary Outcome: Proportion of Subjects Achieving Undetectable HCV RNA at Week 4 and Week 12
Description: number of subjects with undetectable HCV RNA
Time Frame: 4 and 12 weeks after the first dose of study drug
Population: Subjects who were randomized and received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Part A: T/PR | Part A: Pbo/PR | Part B: EFV-based HAART + T/PR | Part B: EFV-based HAART + Pbo/PR | Part B: ATV/R-based HAART + T/PR | Part B: ATV/R-based HAART + Pbo/PR
Number analyzed (Participants) | 7 | 6 | 16 | 8 | 15 | 8
participants
  Week 4 (RVR) | 5 | 0 | 12 | 0 | 9 | 0
  Weeks 4 and 12 (eRVR) | 4 | 0 | 12 | 0 | 7 | 0

3. Secondary Outcome: Proportion of Subjects Who Have Undetectable HCV RNA 12 Weeks (SVR12) and 24 Weeks (SVR24) After Last Planned Dose of Study Treatment
Time Frame: 12 weeks after last dose of study drug
Population: subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part A: T/PR | Part A: Pbo/PR | Part B: EFV-based HAART + T/PR | Part B: EFV-based HAART + Pbo/PR | Part B: ATV/R-based HAART + T/PR | Part B: ATV/R-based HAART + Pbo/PR
Number analyzed (Participants) | 7 | 6 | 16 | 8 | 15 | 8
participants
  SVR12 | 5 | 2 | 11 | 4 | 12 | 4
  SVR24 | 5 | 2 | 11 | 4 | 12 | 4

4. Secondary Outcome: Effect of Efavirenz-based (EFV) and Atazanavir-based (ATV/r) Highly Active Antiretroviral Therapy(HAART) on Telaprevir Exposure
Time Frame: through 12 weeks after first dose of study drug
Population: subjects with available plasma concentration data
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio (test/reference)
Arm/Group | EFV-based (Test, N=15) vs No HAART (Reference, N=7) | ATV/R-based (Test, N=13) vs No HAART (Reference, N=7)
Number analyzed (Participants) | 15 | 13
ratio (test/reference)
  Cmin | 0.8842 [0.5467 to 1.4300] | 1.3059 [0.7981 to 2.1367]
  Cavg | 0.9610 [0.6615 to 1.3961] | 1.0930 [0.7456 to 1.6023]
  Cmax | 1.0061 [0.7306 to 1.3855] | 1.0075 [0.7260 to 1.3982]

5. Secondary Outcome: Median Trough Plasma Concentration (Ctrough) Ratios of Efavirenz and Tenofovir (Part B Only, Subjects on EFV-based HAART)
Description: Ctrough ratio of HAART medication with telaprevir (test) and without telaprevir (reference)
Time Frame: through 12 weeks after first dose of study drug
Population: subjects with available concentration data
Measure: Median (Full Range); unit: ratio (test/reference)
Groups:
- T/PR: Telaprevir plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant efavirenz(EFV)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
- Pbo/PR: Placebo plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant efavirenz(EFV)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
Arm/Group | T/PR | Pbo/PR
Number analyzed (Participants) | 14 | 8
ratio (test/reference)
  Efavirenz | 0.94 [0.42 to 2.84] | 0.79 [0.48 to 1.48]
  Tenofovir | 1.06 [0.46 to 17.4] | 0.64 [0.30 to 2.01]

6. Secondary Outcome: Median Trough Plasma Concentration (Ctrough) Ratios of Atazanavir (ATZ), Ritonavir, and Tenofovir (Part B Only, Subjects on ATV-based HAART)
Description: Ctrough of HAART medication with telaprevir (test) and without telaprevir (reference)
Time Frame: through 12 weeks after first dose of study drug
Population: subjects with available concentration data
Measure: Median (Full Range); unit: ratio (test/reference)
Groups:
- T/PR: Telaprevir plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant ritonavir-boosted atazanavir(ATV/r)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
- Pbo/PR: Placebo plus peginterferon alfa-2a and ribavirin for 12 weeks, followed by 36 weeks of peginterferon alfa-2a and ribavirin. Subjects receiving concomitant ritonavir-boosted atazanavir(ATV/r)-based highly active antiretroviral therapy(HAART) for the entire 48 week study.
Arm/Group | T/PR | Pbo/PR
Number analyzed (Participants) | 13 | 7
ratio (test/reference)
  Atazanavir (N=12 T/PR, N=6 Pbo/PR) | 1.16 [0.39 to 45.0] | 1.03 [0.49 to 2.05]
  Tenofovir (N=13 T/PR, N=7 Pbo/PR) | 0.75 [0.28 to 40.7] | 0.93 [0.55 to 1.68]
  Ritonavir (N=9 T/PR, N=7 Pbo/PR) | 0.72 [0.08 to 4.40] | 0.74 [0.21 to 4.20]

ADVERSE EVENTS:
Time Frame: first dose of study drug until 4 weeks after the last dose of study drug
Groups:
- T/PR: Pooled T/PR from Part A and Part B
- Total PR: Pooled PR from Part A and Part B
Arm/Group | T/PR | Total PR
Serious Adverse Events (participants affected / at risk) | 7/38 | 2/22
Other Adverse Events (participants affected / at risk) | 38/38 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T/PR (N=38) | Total PR (N=22)
Groin Infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Cellulitis Staphylococcal (Infections and infestations) | 1 | 0
Staphylococcal Abscess (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hemolytic Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T/PR (N=38) | Total PR (N=22)
Chills (General disorders) | 6 | 4
Pyrexia (General disorders) | 8 | 2
Influenza-like Illness (General disorders) | 5 | 3
Irritability (General disorders) | 5 | 3
Fatigue (General disorders) | 16 | 9
Injection Site Erythema (General disorders) | 2 | 1
Pain (General disorders) | 1 | 3
Malaise (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 13 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 4
Vomiting (Gastrointestinal disorders) | 7 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 3
Anogenital Dysplasia (Gastrointestinal disorders) | 0 | 2
Cheilitis (Eye disorders) | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Headache (Nervous system disorders) | 14 | 6
Dizziness (Nervous system disorders) | 8 | 3
Paraesthesia (Nervous system disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2
Depression (Psychiatric disorders) | 8 | 2
Insomnia (Psychiatric disorders) | 5 | 5
Anxiety (Psychiatric disorders) | 3 | 1
Depressed Mood (Psychiatric disorders) | 1 | 3
Affect Lability (Psychiatric disorders) | 2 | 0
Libido Decreased (Psychiatric disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Fungal Skin Infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 5
Anaemia (Blood and lymphatic system disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Weight Decreased (Investigations) | 5 | 5
Blood Bilirubin Increased (Investigations) | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days